CLINICAL TRIAL: NCT06417853
Title: Phase I Clinical Study to Evaluate the Safety and Tolerability of a Monovalent Influenza a (H7N9) Vaccine Delivered Intradermally by High-density Microarray Patch (HD-MAP) in Healthy Adults Aged 18 to 50 Years
Brief Title: Influenza a (H7N9) Vaccine Delivered Intradermally by High-density Microarray Patch (HD-MAP)
Acronym: HD-MAP
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxxas Pty Ltd (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SP-1219-007
Record Dates: First submitted 2024-05-08; First posted 2024-05-16 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: H7N9 Influenza
Keywords: Influenza A Monovalent Vaccine Microarray Delivery System
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study will be mixed and will contain open label and double-blinded groups; the active comparator groups (Group 1: H7N9 unadjuvanted IM and Group 4: H7N9 with MF59® IM) will be open-label whilst groups (Groups 2, 3 and 5 to 8: VXS-1219 and VXS-1219A) will be double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Arm 1: Influenza A (H7N9) Vaccine Intramuscular Injection (Active Comparator): 7.5 mcg HA unadjuvanted IM injection (n=30)
- Arm 2: Unadjuvanted Influenza A (H7N9) Vaccine Microarray Patch (Experimental): VXS-1219 12 mcg HA (n=30) and VXS-1219U (n =3)
  Interventions: Combination Product: Unadjuvanted Influenza A (H7N9) Monovalent Vaccine Microarray Patch Delivery System (low dose HA); Device: Microarray Patch Delivery System
- Arm 3: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch (Experimental): VXS-1219 25 mcg HA (n=30) and VXS-1219U (n =3)
  Interventions: Combination Product: Adjuvanted Influenza A (H7N9) Monovalent Vaccine Microarray Patch Delivery System (high dose HA); Device: Microarray Patch Delivery System
- Arm 4: Adjuvanted Influenza A (H7N9) Vaccine Intramuscular Injection (Active Comparator): 7.5 mcg HA with MF59® adjuvant 7.5 IM injection (n=30)
  Interventions: Biological: Adjuvanted Influenza A (H7N9) Monovalent Vaccine Injection
- Arm 5: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch (Experimental): VXS-1219A 12 mcg HA + QS21 4 mcg (n=30) and VXS-1219U (n =3)
  Interventions: Combination Product: Adjuvanted Influenza A (H7N9) Monovalent Vaccine Microarray Patch Delivery System (low dose HA, low dose adjuvant); Device: Microarray Patch Delivery System
- Arm 6: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch (Experimental): VXS-1219A 12 mcg HA + QS21 8 mcg (n=30) and VXS-1219 (n = 3)
  Interventions: Combination Product: Adjuvanted Influenza A (H7N9) Monovalent Vaccine Microarray Patch Delivery System (low dose HA, high dose adjuvant); Device: Microarray Patch Delivery System
- Arm 7: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch (Experimental): VXS-1219A 20 mcg HA + QS21 3.3 mcg (n=30) and VXS-1219U (n=3)
  Interventions: Combination Product: Adjuvanted Influenza A (H7N9) Monovalent Vaccine Microarray Patch Delivery System (high dose HA, low dose adjuvant); Device: Microarray Patch Delivery System
- Arm 8: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch (Experimental): VXS-1219A 20 mcg HA + QS21 6.7 mcg (n=30) and VXS 1219U (n=3)
  Interventions: Combination Product: Adjuvanted Influenza A (H7N9) Monovalent Vaccine Microarray Patch Delivery System (high dose HA, high dose adjuvant); Device: Microarray Patch Delivery System

INTERVENTIONS:
Biological: Unadjuvanted Influenza A (H7N9) Monovalent Vaccine Injection — 7.5 mcg Influenza A (H7N9) Injection
Combination Product: Unadjuvanted Influenza A (H7N9) Monovalent Vaccine Microarray Patch Delivery System (low dose HA) — 12 mcg Influenza A (H7N9) Microarray Patch Delivery System (VXS-1219)
  Arms: Arm 2: Unadjuvanted Influenza A (H7N9) Vaccine Microarray Patch
Combination Product: Adjuvanted Influenza A (H7N9) Monovalent Vaccine Microarray Patch Delivery System (high dose HA) — 25 mcg Influenza A (H7N9) Microarray Patch Delivery System (VXS-1219)
  Arms: Arm 3: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch
Biological: Adjuvanted Influenza A (H7N9) Monovalent Vaccine Injection — 7.5 mcg Influenza A (H7N9) with MF59® Injection
  Arms: Arm 4: Adjuvanted Influenza A (H7N9) Vaccine Intramuscular Injection
Combination Product: Adjuvanted Influenza A (H7N9) Monovalent Vaccine Microarray Patch Delivery System (low dose HA, low dose adjuvant) — 12 mcg Influenza A (H7N9) with 4 mcg QS21 Microarray Patch Delivery System (VXS-1219A)
  Arms: Arm 5: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch
Combination Product: Adjuvanted Influenza A (H7N9) Monovalent Vaccine Microarray Patch Delivery System (low dose HA, high dose adjuvant) — 12 mcg Influenza A (H7N9) with 8 mcg QS21 Microarray Patch Delivery System (VXS-1219A)
  Arms: Arm 6: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch
Combination Product: Adjuvanted Influenza A (H7N9) Monovalent Vaccine Microarray Patch Delivery System (high dose HA, low dose adjuvant) — 20 mcg Influenza A (H7N9) with 3.3 mcg QS21 Microarray Patch Delivery System (VXS-1219A)
  Arms: Arm 7: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch
Combination Product: Adjuvanted Influenza A (H7N9) Monovalent Vaccine Microarray Patch Delivery System (high dose HA, high dose adjuvant) — 20 mcg Influenza A (H7N9) with 6.7 mcg QS21 Microarray Patch Delivery System (VXS-1219A)
  Arms: Arm 8: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch
Device: Microarray Patch Delivery System — Vaccine free Microarray Patch Delivery System (VXS-1219U)
  Arms: Arm 2: Unadjuvanted Influenza A (H7N9) Vaccine Microarray Patch; Arm 3: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch; Arm 5: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch; Arm 6: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch; Arm 7: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch; Arm 8: Adjuvanted Influenza A (H7N9) Vaccine Microarray Patch

SUMMARY:
Study SP-1219-007 is a multi-centre, randomised, study designed to access the safety and tolerability of two doses of monovalent Influenza A (H7N9) vaccine delivered intradermally by a microarray patch delivery system in healthy adults aged 18 to 50 years.

DETAILED DESCRIPTION:
258 participants will be randomized to receive two doses (Day 1 and 22) of either VXS-1219, VXS-1219 with QS21 adjuvant (VXS-1219A), an intramuscular comparator (H7N9 vaccine or H7N9 + MF59® vaccine) or an uncoated, vaccine-free HD-MAP Delivery system (VXS-1219U). VXS-1219A is identical to VXS-1219 with the only difference being this investigational product will be formulated with QS21. VXS-1219U, the vaccine-free microarray patch delivery system comparator, includes a terminally sterilized polymer patch and does not include any vaccine coating formulation on the micro-projections, but is otherwise identical to VXS-1219 and VXS-1219A.

The primary objective of the study is to evaluate the safety and tolerability of two doses of H7N9 Influenza A vaccine (12 to 25 mcg HA) with and without QS21 adjuvant (3.3 to 8 mcg), administered by the microarray patch delivery system, compared to IM H7N9 vaccine (7.5 mcg HA) with and without MF59® and uncoated, vaccine-free microarray patch delivery system, administered 21 days apart.

The secondary objectives of the study are to evaluate the immune response to two doses H7N9 Influenza A vaccine (12 to 25 mcg HA) with and without QS21 adjuvant (3.3 to 8 mcg), administered by the microarray patch delivery system, compared to IM H7N9 vaccine (7.5 mcg HA) with and without MF59® and uncoated, vaccine-free microarray patch delivery system, administered 21 days apart.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria to be eligible for this study:

* Aged 18 to 50 years (inclusive) at the time of consent;
* Body mass index (BMI) within the range 18.0 to 32.0 kg/m² (inclusive) at Screening;
* Being in good health, as determined by satisfactory physical examination, vital signs, 12-lead ECG, laboratory evaluation, stable medical history and clinical judgment of the Investigator. Participants with stable, chronic underlying illnesses such as psychiatric/psychological disorders, hypertension, diabetes, ischemic heart disease or hypothyroidism (or other conditions as per investigator's discretion) may be enrolled at the discretion of the PI and provided their signs and symptoms are controlled. If on regular prescription medication, the medication dose must have been stable for at least three months prior to Screening;
* Adequate venous access in left or right arm to allow collection of small-volume blood samples at different visits;
* Participants of childbearing potential must return a negative pregnancy test at Screening (serum) and pre-dose on Day 1 (urine), and must agree to remain sexually abstinent, use medically effective contraception or have a partner who is sterile or same-sex, from Screening through to Day 78. The use of medically effective contraception or IUD must be stable for at least three months prior to Screening. Surgical sterilisation, e.g., tubal ligation, hysterectomy and bilateral oophorectomy in women, or vasectomy in men, is required at least six months prior to Screening. Post menopausal participants can be included, and are defined as those with at least 12 months since their last menstrual period;
* Non-surgically sterilised, sexually active male participants with a female partner of child-bearing potential must agree to use condoms, together with medically effective contraception for their female partner through to Day 78;
* Participant is able to communicate effectively with study personnel and is considered likely to be reliable, willing and cooperative in terms of compliance with the protocol requirements;
* Participant is able and willing to provide written, personally signed, informed consent to participate in the study

Exclusion Criteria:

Participants meeting any of the following exclusion criteria will not be eligible for this study:

* Participants who have received any registered vaccine within 30 days prior to Day 1;
* Planned administration of any registered vaccine prior to the immunogenicity blood draw on Day 43;
* Previous administration of any H7 vaccine, previous physician-confirmed H7 disease, previous known or potential exposure to avian influenza virus H7N9 HA antigen or any other avian influenza including H5N1, at any time in the past;
* Participants with birthmarks, tattoos, wounds, scars, moles, blemishes, heavy hair or other skin conditions (such as eczema) at the planned vaccination sites (2 adjacent sites overlying the deltoid muscle which are at least 3 cm apart) that could be expected to obscure the observation of treatment site reactions. If dosing on Day 22 is performed on different arm than Day 1, the same exclusion criteria shall apply;
* Participant with known chronic spontaneous urticaria or dermographism;
* Known predisposition to keloid-scar formation (participants who have developed a scar caused by BCG vaccine can be included in the study);
* Known anaphylactic hypersensitivity to haemagglutinin or to any of the vaccine or adjuvant excipients (squalene, polysorbate 80, sorbitan trioleate, sodium citrate dihydrate, citric acid monohydrate, protein other than H7N9 including Madin Darby Canine Kidney (MDCK) cell protein, (residual), MDCK cell DNA, (residual), cetyltrimethylammonium bromide (residual), beta-propiolactone (residual), QS21 extract, or any other excipient contained in the study products;
* Allergy to a previous vaccination at any time in the past;
* Known history of demyelinating disease or Guillain-Barré syndrome;
* History of granulomatous diseases, including sarcoidosis and granuloma annulare;
* History of convulsions, epilepsy, other physician diagnosed central nervous system diseases, excluding febrile convulsions experienced as a child that are considered resolved;
* History of clinically significant haematological, gastrointestinal, hepatic, renal, cardiovascular, dermatological, immunological, respiratory, endocrine, oncological, neurological, metabolic, psychiatric disease, that, at the discretion of the Investigator, precludes the participant from the study;
* Presence of active viral or bacterial infection, with or without fever (tympanic temperature ≥38.0 °C), at Day 1 or within 72 hours prior to study vaccination, if determined by the Investigator to be of clinical significance. Participants with a minor illness such as mild diarrhoea or mild upper respiratory infection without fever may be enrolled at the discretion of the Investigator. Enrolment may be deferred for up to one week provided participant remains otherwise eligible and the total Screening period does not exceed 14 days;
* History of any haematological malignancy or active neoplastic disease (Non-melanoma skin cancer that was successfully treated within the 5 year period can be included in the study). Active is defined as having received treatment within the five years prior to Screening;
* Presence of an active medical condition, defined as a condition under current evaluation or treatment, that is considered clinically significant by the Investigator, or a recent illness that is considered clinically significant by the Investigator;
* Any condition that, in the opinion of the Investigator, is considered clinically significant or might interfere with the evaluation of the study objectives;
* Planned surgery requiring a general anaesthetic, or surgery requiring inpatient hospitalisation for at least 24 hours from Screening through to Day 78;
* History of illness and/or infection with Hepatitis B, or Hepatitis C or Human Immunodeficiency Virus (HIV), or a positive test for Hepatitis B surface antigen, Hepatitis C or antibodies against HIV at Screening;
* History of abnormal bleeding, and/or thrombophlebitis unrelated to venepuncture or intravenous cannulation;
* History of autoimmune or autoinflammatory immune-mediated medical conditions;
* Receiving chronic treatment with immunosuppressive therapy, including chronic use (more than 14 continuous days) of corticosteroids within 30 days prior to Day 1.
* Participant who has received immunoglobulins and/or any blood or blood products within three months prior to Day 1 or plans to receive any blood or blood products at any time during the study;
* Participant who has donated blood or plasma, or has had clinically significant blood loss, within 14 days prior to Day 1. Participants who plan to donate blood or plasma within 12 weeks of dose 2 should also be excluded;
* Female participant who is pregnant or breast-feeding, or intends to become pregnant, from Screening through EoS;
* A history of alcohol or drug abuse in the past 12 months, or current declared alcohol consumption >4 standard drinks per day for 7 days per week (one standard drink is equivalent to 285 mL of full-strength beer, 100 mL of wine or 30 mL of spirits);
* Use of any prescription medication (with the exception of contraceptives, hormone replacement therapy, or stable doses of medication required for the management of stable, chronic underlying illnesses) within seven days prior to Day 1;
* Use of any investigational drug or device within 30 days, or five half-lives of the drug (whichever is longer) before Day 1, or planned use of another investigational drug or device at any time during the study;
* An employee, or a first-degree family member of an employee, of the Sponsor, Contract Research Organization conducting this study, or study site involved in this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 267 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and duration of solicited systemic adverse reactions including fever, headache, malaise, myalgia, arthralgia, fatigue, sweating and shivering from Day 1 through Day 8 (Dose 1) and Day 22 through Day 29 (Dose 2); | 387 days
Incidence, severity and duration of local adverse reactions including erythema, swelling, induration, ecchymosis, and vaccination site pain from Day 1 through Day 8 (Dose 1) and Day 22 through Day 29 (Dose 2); | 387 days
Incidence and severity of unsolicited (spontaneously reported) treatment-emergent adverse events (TEAEs) from Day 1 through Day 78; | 78 days
Incidence and severity of SAEs, MAAEs and PIMMCs from Day 1 through Day 387; | 387 days
Incidence and severity of Application Site Reactogenicity Adverse Events with onset after Day 78 from Day 79 through Day 387; | 387 days
Number of Participants with Clinically Significant Changes in Laboratory Tests from Day 1 to Day 387; | 387 days
  Clinical safety laboratory tests include Hematology, Biochemistry panel, Serology for Hepatitis B and C (HBsAg, HCV) and HIV (HIV-1 and HIV-2), Beta-human chorionic gonadotropin (HCG) serum pregnancy test for female participants of childbearing potential only. Females with natural amenorrhea for <12 months and who ate not surgically sterile, and Urine pregnancy dipstick test will be performed onsite at pre-dose Day 1 and pre dose Day 22 for female participants of childbearing potential only.
Number of Participants with Clinically Significant Changes in Physical Examination from Day 1 to Day 387 | 387 days
  A complete physical examination will include assessments of general appearance; skin and lymphatics; head; eyes; ears; nose; throat; cardiovascular system; respiratory system; abdomen/gastrointestinal system; musculoskeletal and neurological systems. Other body systems may also be examined as required, at the discretion of the Investigator.
Number of Participants with Clinically Significant Changes in Vital Signs from Day 1 through Day 387; | 387 days
  Vital sign measurements will include tympanic body temperature (in degrees Celsius [°C]), systolic and diastolic blood pressure (in millimeters of mercury [mmHg]), heart rate (in beats per minute) and respiratory rate (number of breaths per minute).
Local skin response, assessed by photo imaging and standardised scoring, measured at 10 minutes and 1 hour following application on Day 1 and Day 22, and at Days 4, 8, 29, and 78; | 78 days
Concomitant medication usage. | 387 days

SECONDARY OUTCOMES:
GMT of serum antibody response to H7N9 antigen, assessed by hemagglutination inhibition assay (HAI) at baseline and Days 8, 22, 29, 43, 78 and 387; | 387 days
GMT of the serum virus neutralising antibody titres to H7N9 antigen, assessed by microneutralisation (MN) assay at baseline and Days 8, 22, 29, 43, 78 and 387. | 387 days
GMT of serum antibody response to H7N9 antigen, seroconversion rate and % of subjects seropositive, assessed by hemagglutination inhibition assay (HAI) at baseline and Days 8, 22, 29, 43, 78 and 387. | 387 days
Seroconversion based on serum HAI antibody titres, defined as either a pre-vaccination HAI titre < 1:10 and a post-vaccination HAI titre ≥ 1:40, or a pre-vaccination HAI titre ≥ 1:10 and a minimum 4-fold increase in post-vaccination HAI titre. | 387 days

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - University of Sunshine Coast Clinical Trials, Morayfield, Queensland
  - University of Sunshine Coast Clinical Trials, Sippy Downs, Queensland
  - University of Sunshine Coast Clinical Trials, South Brisbane, Queensland
  - Doherty Clinical Trials Ltd, East Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No